

# **CLINICAL STUDY PROTOCOL**

Title: A Prospective, Multi-Center Study of Phasix<sup>TM</sup> Mesh for

Ventral or Incisional Hernia Repair.

Protocol Number: DVL-HE-011

Study Type: Post-market, multi-center, prospective, open label

**Date:** October 30, 2017

Version: 4.0

Study Devices: Phasix<sup>TM</sup> Mesh

Sponsor: Davol Inc.

Subsidiary of C. R. Bard, Inc. 100 Crossings Boulevard Warwick, RI 02886 Phone: 1-800-556-6756

**Sponsor Contacts:** Rushil Sankpal

**Project Manager, Corporate Clinical Affairs** 

C. R. Bard, Inc. 730 Central Avenue Murray Hill, NJ 07974 Telephone: 908-277-8082

Email: Rushil.sankpal@crbard.com

## **Protocol Signature Page**

The Investigator agrees to conduct the clinical study, which is the subject of this protocol, in accordance with the Clinical Study Agreement, this protocol, all applicable laws and regulations, and the conditions of approval imposed by the reviewing Institutional Review Board.

| Agreed to by (Investigator): |
|------------------------------|
| Printed Name – Investigator |
| Signature – Investigator |
| Date |

# **Protocol Abbreviations/Acronyms**

| Abbreviation/Acronym | Definition |
|----------------------|-----------------------------------------------------|
| AE | Adverse event |
| Bard | C. R. Bard, Inc. |
| BMI | Body Mass Index |
| CDC | US Centers for Disease Control and Prevention |
| CFR | Code of Federal Regulations |
| Cm | Centimeter |
| CT | Computed Tomography Scan |
| COPD | Chronic Obstructive Pulmonary Disease |
| CST | Component Separation Technique |
| CV | Curriculum vitae |
| eCRF | Electronic Case Report Form |
| e.g. | For Example |
| FDA | Food and Drug Administration |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human Immunodeficiency Virus |
| Hrs | Hours |
| ICF | Informed Consent Form |
| i.e. | That Is |
| IRB | Institutional Review Board |
| IFU | Instructions For Use |
| LTF | Lost to Follow-Up |
| Mm | Millimeter |
| MRI | Magnetic Resonance Imaging |
| N | Sample Size |
| P4HB | poly-4-hydroxybutyrate |
| PE | Physical Exam |
| SAE | Serious Adverse Event |
| SF-12® | 12-Item Short Form |
| SSI | Surgical Site Infection |
| VAC | Vacuum Assisted Closure system |
| VAS | Visual Analogue Scale |

## **TABLE OF CONTENTS**

| 1 | | INTRODUCTION | 7 |
|---|-------|-------------------------------------------|------|
| | 1.1 | Background | 7 |
| | 1.2 | Rationale | 9 |
| | 1.3 | Device Descriptions | 9 |
| | 1.3.1 | Phasix <sup>TM</sup> Mesh | 9 |
| 2 | | STUDY OBJECTIVES | 9 |
| 3 | | STUDY ENDPOINTS | 9 |
| 4 | | STUDY DESIGN | . 10 |
| 5 | | STUDY POPULATION | . 11 |
| | 5.1 | Number Of Subjects | . 11 |
| | 5.2 | Eligibility Criteria – Enrollment Period | . 11 |
| | 5.2.1 | Inclusion Criteria | . 11 |
| | 5.2.2 | Exclusion Criteria | . 11 |
| | 5.3 | Eligibility Criteria – Extension | . 12 |
| | 5.3.1 | Inclusion Criteria | . 12 |
| | 5.3.2 | Exclusion Criteria | . 12 |
| 6 | | STUDY PROCEDURES | . 12 |
| | 6.1 | Subject Screening and Baseline Evaluation | . 12 |
| | 6.1.1 | Informed Consent. | . 13 |
| | 6.1.2 | Enrollment | . 13 |
| | 6.1.3 | Eligibility | . 13 |
| | 6.1.4 | Assignment of Subject Screening Number | . 14 |
| | 6.1.5 | Blinding | . 14 |
| | 6.1.6 | Demographics and Medical History | . 14 |
| | 6.1.7 | Physical Examination | . 14 |
| | 6.1.8 | Concomitant Pain Medication Usage | . 14 |
| | 6.1.9 | Patient Reported Outcome Assessments | . 14 |
| | 6.2 | Surgical Procedure | . 14 |
| | 6.2.1 | General Procedures | . 14 |
| | 6.2.2 | Component Separation Technique Surgery | . 15 |

| ctober 30, 2017 |
|-----------------|
| 15 |
| 16 |

| 12 | .2 | Investigator Selection | 28 |
|----|------|---------------------------------------------|----|
| 12 | .3 | Regulatory and Ethical Considerations | 28 |
| | 12.3 | .1 Institutional Review Board Approval | 29 |
| | 12.3 | .2 Informed Consent and HIPAA Authorization | 29 |
| | 12.3 | .3 Confidentiality | 29 |
| 12 | .4 | Protocol Adherence and Deviations | 29 |
| 12 | .5 | Device Accountability | 30 |
| 12 | .6 | Data Collection | 30 |
| 12 | .7 | Subject Compensation | 30 |
| 12 | .8 | Communications with the Sponsor | 30 |
| 12 | .9 | Required Documentation | 30 |
| 13 | | SITE MONITORING | 31 |
| 13 | .1 | Study Initiation Visit | 31 |
| 13 | .2 | Ongoing Monitoring Visits | 33 |
| 13 | .3 | Final Monitoring Visit | 33 |
| 14 | | TERMINATION OF STUDY | 33 |
| 15 | | REPORTING REQUIREMENTS | 33 |
| 16 | | RECORD RETENTION | 34 |
| 17 | | REFERENCES | 35 |
| 18 | | APPENDICES | 38 |

#### 1 INTRODUCTION

## 1.1 Background

With more than 2 million abdominal operations occurring annually in the United States (US), up to 20% of those patients developing ventral incisional hernias, abdominal wall defects and incisional hernias represent a challenging surgical condition. Approximately 250,000 ventral hernia repairs are performed on a yearly basis. There are several options for repair, including primary repair, synthetic or biologic material placement, repair with relaxing incisions, and use of musculofascial flaps, utilizing both open and laparoscopic approaches. However, there is no clear-cut consensus regarding the optimal hernia repair technique, particularly in complex hernia repair cases where patient co-morbidities exist and a high risk of infection is present.

Simple suture repair has been associated with a high risk of hernia recurrence, with reports ranging from 10% to 55%, and has been nearly abandoned for the repair of hernias which are greater than five centimeters (cm) in size.<sup>4, 5, 6, 7</sup> As a result, many ventral hernia repair procedures involve the use of a mesh material.

Synthetic mesh repair procedures, either open or laparoscopic, have been reported to lead to fewer recurrences compared to primary repairs. <sup>8, 9, 10</sup> Improved outcomes are believed to be related to reduced tension on the fascial edges and sutures when mesh is used in hernia repair procedures. However, complex cases and large abdominal wall defects continue to pose a challenge to surgeons. Factors such as patient co-morbidities, defect size, location, tissue viability and degree of contamination are included in a surgeon's assessment and decision-making process. <sup>11</sup> These large abdominal wall defects have been associated with recurrence rates of up to 46%. <sup>12</sup>

Despite reducing hernia recurrence rates, the use of synthetic mesh has been associated with complications such as infection, adhesions, fistulae, and foreign body reactions including increased inflammation and/or connective tissue deposition.<sup>13</sup>

Non-absorbable meshes can lead to complications related to the body's reaction to the persistent foreign mesh material resulting in foreign body sensations including discomfort and chronic pain, which is described by the International Association for the Study of Pain as pain lasting for 3 months or greater following hernia repair. 14, 15

Ideally, an absorbable mesh would provide adequate structural support throughout the healing process and would be fully absorbed when the wound has completely healed, thereby potentially reducing the chances for complications associated with the persistence of non-absorbable mesh material. However, the development of absorbable mesh products has faced challenges related to the rate of absorption with complications arising when the mesh product is absorbed too quickly. Rapid absorption does not support sufficient healing if structural reinforcement is diminished during the tissue repair period. An absorbable mesh should

Davol Inc. Version 4.0 Phasix $^{TM}$  Mesh October 30, 2017 Protocol DVL-HE-011

retain its functional strength for a sufficient period of time to allow native cellular ingrowth tissue remodeling, maturation of collagen, and gradual shift of mechanical load.

Phasix<sup>TM</sup> Mesh is a commercially available medical device in the US. It is a resorbable mesh prepared from poly-4-hydroxybutrate (P4HB) which has been studied for use as a biomaterial for a number of applications in medical devices and tissue engineering due to favorable mechanical properties, biocompatibility and desirable degradation times. <sup>16, 17, 18</sup> Using standard measures of mechanical strength (suture pull-out, tear and ball burst strength) Phasix<sup>TM</sup> Mesh is comparable in performance to traditional polypropylene mesh. Pre-clinical implantation studies indicate that the resorption of the Phasix<sup>TM</sup> Mesh fibers is minimal throughout the 12 week expected period of healing and up to ~26 weeks post-implantation. Resorption of the fibers is essentially complete in 12-18 months. <sup>19, 20</sup> Given the long-term strength retention observed in preclinical studies, it is anticipated that Phasix<sup>TM</sup> Mesh may result in low recurrence and complication rates with minimal pain and discomfort when used for hernia repair.

A porcine bridging hernia repair study demonstrated that Phasix<sup>TM</sup> Mesh could perform as a durable scaffold for soft tissue repair when spanning a surgical defect.<sup>20</sup> The results of the 52-week study showed that the repair site had significantly greater mechanical repair strength, as compared to native abdominal wall. This persisted even after significant Phasix<sup>TM</sup> Mesh resorption (as measured by molecular weight). Phasix<sup>TM</sup> Mesh showed an initial mild-moderate host inflammatory response, that declined to mild over 52 weeks. Neovascularization (angiogenesis) and new collagen deposition were evident at 6, 12, 26 and 52 weeks. In a 24-week rat study, histological analyses of the repair site demonstrated that some competitive meshes had a greater overall host inflammatory response, some had less of a response and one had a very similar response, to Phasix<sup>TM</sup> Mesh.<sup>21</sup> In the same study, histological analyses demonstrated similar variability on measures of host fibrotic response.

MonoMax<sup>®</sup> suture (B. Braun Melsungen AG) is a product made from the same polymer as Phasix<sup>TM</sup> Mesh. A twelve month, 150-patient, multicenter clinical study demonstrated the safety and efficacy of MonoMax<sup>®</sup> for abdominal wall closure.<sup>22</sup> Wound infection and wound dehiscence rates were compared between MonoMax<sup>®</sup> and an historical control (7.3% versus 11.3% combined). One year after surgery, the rate of incisional hernias was similar comparing the two groups: 21 patients (14.0%) in the MonoMax<sup>®</sup> group compared to 30 patients (21.3%) in the control.

This post-approval clinical study is being conducted to evaluate the use of Phasix<sup>™</sup> Mesh in primary ventral, incisional or multiply-recurrent hernia repair in patients with a higher level of risk as defined by the presence of 1 or more common pre-existing conditions. Patients who receive a Phasix<sup>™</sup> Mesh implant will be followed for 60 months.

#### 1.2 Rationale

This study is intended to evaluate the use of Phasix<sup>TM</sup> Mesh for primary ventral, incisional and multiply-recurrent incisional hernia repair amongst subjects at high risk for complications. This protocol version (4.0) is intended to capture longer term data (through 60 months) on all eligible subjects. The protocol's follow up period was not extended due to safety related concerns or trends.

## 1.3 **Device Descriptions**

#### 1.3.1 Phasix<sup>TM</sup> Mesh

The Phasix<sup>TM</sup> Mesh (Davol, Inc.) is a resorbable mesh prepared from P4HB. P4HB is produced from a naturally occurring monomer and is processed into monofilament fibers and knitted into a surgical mesh. Phasix<sup>TM</sup> Mesh degrades through a process of hydrolysis and a hydrolytic enzymatic digestive process. It was developed to minimize the variability of resorption rate (loss of mass) and strength and provide support throughout the expected period of healing.

Pre-clinical implantation studies indicate that the resorption of the Phasix<sup>TM</sup> fibers is minimal throughout the 12-week expected period of healing and up to about 26 weeks post implantation. Resorption of the fibers is essentially complete in 12 to 18 months. <sup>19, 20</sup>

Phasix<sup>TM</sup> Mesh has been commercially available in the US since 2012 and is indicated to reinforce soft tissue where weakness exists, such as the repair of hernia or other fascial defects that require reinforcement or bridging material to obtain the desired surgical result. Because Phasix<sup>TM</sup> Mesh is fully resorbable, it should not be used in repairs where permanent wound or organ support from the mesh is required. A full description of Phasix<sup>TM</sup> Mesh is included in the product's Instructions for Use (IFU) (Appendix 2).

## 2 STUDY OBJECTIVES

The objective of this study is to collect additional data on safety, performance and effectiveness of Phasix<sup>TM</sup> Mesh in subjects requiring primary ventral, incisional or multiply-recurrent hernia repair in subjects at high risk for complications. Subjects at high risk are defined as having 1 or more of the following co-morbidity conditions: body mass index (BMI) between 30-40 kg/m², inclusive, active smokers, chronic obstructive pulmonary disease (COPD), diabetes, immunosuppression, coronary artery disease, chronic corticosteroid use, low pre-operative serum albumin, advanced age, or renal insufficiency. The study end points are described below.

#### 3 STUDY ENDPOINTS

There are two primary endpoints, hernia recurrence rate and surgical site infection (SSI) rate, and six secondary endpoints:

## 3.1 Primary Endpoints:

#### 1. Hernia Recurrence Rate

Hernia recurrence rates will be assessed by physical examination at each study visit through 60 months. A recurrent hernia will be defined as any hernia identified or confirmed by the investigator, during any study follow-up visit, in approximately the same position as the hernia repaired in the study procedure. Potential hernias identified via incidental magnetic resonance imaging (MRI) or computed tomography (CT) scan will be evaluated by the operating surgeon for clinical significance and confirmation of hernia recurrence.

## 2. Surgical Site Infections

Infections at the surgical site will be assessed by physical examination at each study visit through 60 months. If an infection is suspected, a routine culture, obtained via each site's standard protocol, should be obtained to determine cell count and type (i.e. yeast, gram positive or gram negative bacteria, or other). If genus and species of the culture are identified as part of the routine practice at the site, that information should be recorded. Classification will follow the CDC guidelines for superficial and deep surgical site infections (Appendix 3).

## 3.2 Secondary Endpoints:

- 1. Pain Visual Analog Scale (VAS)
- 2. Device related adverse event incidence
- 3. Rate of reoperation due to the index hernia repair
- 4. Quality of life assessments (Carolinas Comfort Scale® and SF-12® 12-item short form health survey)
- 5. Surgical procedure time as measured from incision to closure (skin to skin)
- 6. Length of stay

#### 4 STUDY DESIGN

This is a prospective, multi-center open-label study designed to collect additional data on safety, performance and effectiveness of Phasix<sup>TM</sup> Mesh for primary ventral or incisional or multiply-recurrent hernia repair. Follow-up visits will be conducted at 1, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months following surgery. See Section 6 for a detailed schedule of study visits and procedures.

#### 5 STUDY POPULATION

## 5.1 Number Of Subjects

This study is projected to enroll up to 120 subjects at approximately 16 US sites.

## 5.2 Eligibility Criteria – Enrollment Period

#### 5.2.1 Inclusion Criteria

The subject must meet all of the criteria listed below to be enrolled in the study:

- 1. Subject must be 18 years of age or older
- 2. Subject or subject's legally authorized representative must be willing to give written informed consent
- 3. Subject must be diagnosed with primary ventral, incisional hernia or multiply-recurrent (not to exceed 3 recurrences) ventral or incisional hernia
- 4. Subject must have a hernia greater than  $10 \text{ cm}^2$  and  $\leq 350 \text{ cm}^2$
- 5. Subject must be willing to undergo initial ventral, incisional or multiply-recurrent incisional hernia repair using retro-rectus or onlay placement (using absorbable suture) with or without Component Separation Technique (CST)
- 6. Subject is expected to meet the criteria for a Class I wound as defined by the CDC (Appendix 4)
- 7. Subjects must have 1 or more of the following pre-study conditions:
  - a. Body Mass Index (BMI) between 30-40 kg/m<sup>2</sup>, inclusive
  - b. Active smokers (if attempts to quit smoking within two weeks of surgery have failed and the patient is still an active smoker at the time of surgery)
  - c. COPD presence on patient self-report
  - d. Diabetes mellitus
  - e. Immunosuppression
  - f. Coronary Artery Disease
  - g. Chronic corticosteroid use: greater than 6 months systemic use
  - h. Serum albumin less than 3.4 g/dL
  - i. Advanced age: 75 years or older
  - j. Renal insufficiency, defined as serum creatinine concentration ≥2.5 mg/dL

#### 5.2.2 Exclusion Criteria

The subject must be excluded from study enrollment if any of the following criteria are met:

- 1. Subject has had 4 or more previous hernia repairs (of the index hernia)
- 2. The subject has peritonitis
- 3. The subject is on or suspected to be placed on chemotherapy medications during any part of the study
- 4. The subject's Body Mass Index (BMI) is greater than 40 kg/m<sup>2</sup>

- 5. The subject has cirrhosis of the liver and/or ascites
- 6. Subject is American Society of Anesthesiology Class 4 or 5
- 7. Subject is known to be infected with human immunodeficiency virus (HIV)
- 8. Subject has a life expectancy of less than 2 years at the time of enrollment
- 9. Subject has any condition that, in the opinion of the Investigator, would preclude the use of the study device, or preclude the subject from completing the follow-up requirements
- 10. Subject's hernia repair utilizes intra-abdominal mesh placement
- 11. Subject has a surgical wound classified as Class II (Clean-Contaminated), Class III (Contaminated) or Class IV (Dirty-Contaminated) as defined by the CDC (Appendix 4)
- 12. Subject has an active or latent systemic infection
- 13. Subject requires surgical bridge repair as the sole repair
- 14. Subject is pregnant or has plans to become pregnant during the study period or is currently breastfeeding
- 15. Subject has enrolled in another clinical study within the last 30 days
- 16. Subject is part of the site personnel directly involved with this study
- 17. Subject has a known allergy to the test device or component materials (patients with known allergies to tetracycline hydrochloride or kanamycin sulfate should be avoided).

## 5.3 Eligibility Criteria – Extension

#### 5.3.1 Inclusion Criteria

The subject must meet the criteria listed below to be enrolled in the study:

1. Subject or subject's legally authorized representative must be willing to give written informed consent

### 5.3.2 Exclusion Criteria

The subject must be excluded from study enrollment if any of the following criteria are met:

1. Abdominal surgeries where the index procedure site was cut through

#### 6 STUDY PROCEDURES

#### 6.1 Subject Screening and Baseline Evaluation

Subjects with a diagnosis of a primary ventral or incisional hernia or multiply-recurrent hernia requiring surgical repair to close the defect will be screened for potential eligibility against the study protocol inclusion and exclusion criteria, utilizing ordinary standard of care

procedures (e.g. physical examination, blood work, medical evaluation) within 30 days of the date of consent. This may include a full anesthetic work-up customary for hernia repair procedures. Any other standard of care examination or evaluation within 30 days of the date of consent may be considered baseline for study purposes. Prior medical records documenting these tests, examinations and evaluations may be used as the source documents for the baseline visit

During the screening and recruitment process, the Investigator will be responsible for describing the nature of the clinical study, verifying that the eligibility criteria have been met, and obtaining informed consent. Written informed consent and a Health Insurance Portability and Accountability Act (HIPAA) waiver must be obtained prior to performance of any protocol specific procedures.

The following screening/baseline procedures will be conducted and documented.

#### 6.1.1 Informed Consent

The investigator will explain the study to the subject, answer all of the subject's questions, and obtain written informed consent in a language in which the subject is fluent before the collection of any study data or performance of any study procedures.

The subject (or subject's legally authorized representative) must be willing and able to sign and date the informed consent form (ICF) prior to the collection of study data or performance of any study procedures. The original, signed informed consent will be retained with the subjects' records and a copy provided to the subject.

#### 6.1.2 Enrollment

Subjects who sign an informed consent will be considered enrolled in this study. Subjects who provide consent for participation but do not meet all of the study eligibility criteria and do not receive the test device will be considered screen failures.

#### 6.1.3 Eligibility

The subject's eligibility for study enrollment will be reviewed and documented on the appropriate eCRF. At the time of screening, a related progress note must be entered in the source documentation to indicate that all eligibility criteria were reviewed and screening results noted. Final eligibility will be determined intraoperatively.

Subjects who fail to meet eligibility criteria should be considered screen failures and treated according to the Investigator's standard of care. Data are to be collected for screen failure subjects from the time the ICF is signed until the subject is deemed a failure. At a minimum, subject demographics and the reason for failure must be collected; adverse events (AEs) will also be collected and followed through satisfactory resolution or stabilization.

## 6.1.4 Assignment of Subject Screening Number

Subject numbers will be assigned in sequential order, consisting of six digits where the first three digits designate the study site and the last three digits designate the subject number (i.e., subject number 101 001 will be the first subject at site 1; 101 002 will be the second subject at site 1, etc.).

## 6.1.5 Blinding

The study is an open-label study with a single treatment condition. Subjects, investigator (and surgeon) will be not be blinded to the study treatment.

## 6.1.6 Demographics and Medical History

The subject's medical history and demographic information will be documented on the appropriate eCRF. Demographic information will include gender, date of birth, race and ethnicity.

### 6.1.7 Physical Examination

A standard physical exam, appropriate to subjects about to undergo abdominal surgery, will be performed by the physician. Height and weight measurements will be recorded to allow for the calculation of BMI. The subject's ability to participate and meet the follow-up requirements will be established.

## 6.1.8 Concomitant Pain Medication Usage

Prescription and over the counter (OTC) pain medication must be recorded in the source documentation and in the eCRF. All current pain medication will be captured at baseline. Hernia associated pain medication only will be captured at 12, 24, 36, 48, and 60 months.

#### 6.1.9 Patient Reported Outcome Assessments

Subjects will complete the Pain VAS, Carolinas Comfort Scale<sup>®</sup> and SF-12<sup>®</sup> to measure pain, discomfort and quality of life at 1, 3, 6, 12, 18, 24, 36, 48, and 60 months.

## 6.2 Surgical Procedure

#### 6.2.1 General Procedures

All subjects will undergo an open ventral repair of hernias. The size of the hernia is an intraoperative inclusion criterion and must be greater than  $10 \text{ cm}^2$  and  $\leq 350 \text{ cm}^2$ . All other intraoperative exclusion criterion should be verified (e.g., a surgical wound classified as clean-contaminated, contaminated or dirty; absence of an active or latent systemic infection; presence of peritonitis; a hernia bridge as the sole repair procedure). Defect closure must be confirmed

The surgical technique will require retro-rectus or onlay placement (using absorbable suture) with or without Component Separation Technique (CST). Subjects will be administered antibiotics according to hospital protocol.

Subjects are prepared to undergo hernia repair following the instructions supplied by the manufacturers. The IFU for Phasix<sup>TM</sup> Mesh device is presented in Appendix 2.

Phasix<sup>TM</sup> Mesh will be placed in the retro-rectus space with absorbable mesh fixation. The peritoneum should remain posterior to the mesh upon completion of mesh placement. Phasix<sup>TM</sup> Mesh may be cut to shape or size desired for each specific application. To prevent recurrence when repairing hernias, a mesh larger than the defect is required to ensure adequate coverage. The mesh is to be positioned so its edges extend beyond the margins of the defect by at least 5 cm. It is recommended that fixation be placed at approximately 5 to 6 cm intervals (6 to 12 resorbable sutures) around the periphery of the mesh. The edges are then fixated to assure proper closure under correct tension.

The procedure may include CST to obtain site closure. All incisions will be closed with staples and/or sutures and wounds will be dressed with sterile occlusive dressings.

## 6.2.2 Component Separation Technique Surgery

Prophylactic antibiotics will be administered according to hospital protocol. If a prior hernia repair utilizing mesh is in the affected area, every effort should be made to remove any mesh remaining. Once all of the dissection is performed and all of the hernia has been exposed, the largest vertical and transverse dimensions should be recorded.

If the CST is utilized, the surgical technique will be a modification of the "component separation technique" by Ramirez et al. with the graft being implanted into the tissue plane of the surgeon's preference, according to the following: Separation of components may be done via open, posterior or endoscopic/minimally invasive technique as described below.<sup>8, 23</sup>

## 6.2.2.1 Open Technique

After entering the abdominal cavity, adhesiolysis is performed to dissect free any intraabdominal contents from the abdominal wall. The skin and subcutaneous fat are dissected free from the anterior sheath of the rectus abdominal muscle and the external oblique muscle. The external oblique is separated through the aponeurosis approximately 1-3 cm from the edge of the rectus, or through the muscle. If the hernia is subxiphoid in position, release must be done above the rib cage and come across the rectus sheath and muscle at the level of where the pectoralis meets the rectus. The external oblique muscle is separated from the internal oblique muscle, as far laterally as possible (aiming to the anterior axillary line), above and below the hernia by approximately 5 cm.

## 6.2.2.2 Posterior Technique

Posterior component separation with transversus abdominis release (TAR): Starting in the upper third of the abdomen, about 0.5 cm medial to the anterior/posterior rectus sheath junction (linea semilunaris), the posterior rectus sheath is incised to expose the underlying transversus abdominis muscle. The muscle is then divided along its entire medial edge using electrocautery. The use of a right-angled dissector significantly facilitates this release and minimizes injury to the underlying transversalis fascia and peritoneum. Transection of the medial edge of the transversus abdominis muscle allows for entrance to the space between the transversalis fascia and the lateral edge of the divided transversus abdominis muscle. The retromuscular space is bluntly developed further laterally to as far as the lateral border of the psoas muscle to allow for a reinforcement of a visceral sac with a large mesh. Also, if needed, this dissection may be extended superiorly above the costal margin and inferiorly to expose both myopectineal orifices.

## 6.2.2.3 Endoscopic/Minimally Invasive Technique

Make a 2 cm incision in the upper abdomen in a location that is convenient for release (such as directly over the costal margin at the level of the mid clavicular line, or at the tip of the 11<sup>th</sup> rib). Please note: this incision may occasionally need to be placed further lateral to ensure the incision is lateral to the linea semilunaris. Dissect down to the level of the external oblique muscle. Separate the external oblique muscular fibers (this allows for visualization of the underlying internal oblique aponeurosis below). Advance a balloon dissector between the internal and external oblique muscle down to the level of the inguinal ligament. Insufflate the balloon under endoscopic visualization. Remove the dissecting balloon and replace with a trocar (first port). Infuse the lateral abdominal cavity with gas, such as carbon dioxide. Place a second port into the lateral abdominal cavity to allow for dissection. A third port may be used to facilitate easier access to parts of the anatomy. If performing a minimally invasive technique multiple incisions may be used to visualize and release the external oblique under direct visualization. Use cautery or alternatively ultrasonic dissection to divide the external oblique muscle from the costal margin down to the inguinal ligament. Please note: extending the dissection to the level of Scarpa's fascia results in even greater abdominal wall advancement. This technique is generally performed bilaterally.

## 6.2.2.4 Open or Endoscopic Technique

If necessary, resect/debride the edges of the rectus fascia to ensure apposition of healthy well-vascularized tissue as the midline is closed. Care must be taken not to damage the

blood supply and the nerves that run between the internal oblique and transverse muscle and enter the rectus abdominal muscle at the posterior side.

Closure should be performed with permanent or long lasting sutures every 1-2 cm between sutures, for example with an interrupted Figure-8 closure or running stitch. The surgeon should make every effort to close the fascial edges including the use of the component separation technique. If the fascia cannot be closed, the peritoneum of the hernia sac should have been preserved so that this can be closed over the Phasix<sup>TM</sup> to provide vascularized tissue.

If a previous scar of skin is present, the scar should be excised. Scarification products may be used to diminish seroma formation. The fascial and subcutaneous layer should be closed with sutures. The skin should be closed with staples and/or sutures. When skin closure can't be achieved, a wound vac can be used.

## 6.2.3 Postoperative Care

Subjects will be discharged when ambulatory and they have satisfied post anesthesia care criteria. Subjects should be instructed to avoid lifting in excess of ten pounds for six weeks. Early ambulation should be encouraged. Postoperative analgesics will be provided to all subjects. Subjects will be given a prescription for hydrocodone/acetaminophen tablets or an equivalent medication based on local prescribing patterns, medication allergies, and subject needs. Subjects will be instructed to keep the incisions covered and dry for 48 hours after which time the dressing may be removed. Subjects should be instructed to keep the incisions dry except for showers for two weeks. Subjects should also be instructed to call the Investigator for fever in excess of 101°F, redness or swelling at the incisions or surgical site, surgical site drainage, or worsening pain.

If for any reason the mesh is removed and a mesh infection is suspected, routine culture, at the site of the wound, area of contamination, or potential contamination, obtained via each site's normal protocol, should be obtained to determine cell count and type (i.e., yeast, gram positive or gram negative bacteria, or other). If genus and species of the culture are identified as part of the routine practice at the site, that information should be recorded.

## 6.2.4 Surgical Details

Surgical details will be recorded and entered in the appropriate source documentation and eCRF(s). Details will include but may not be limited to procedure date, start/stop times, procedure related complications, and AEs.

#### 6.3 **Subject Follow-up**

Davol Inc. Version 4.0 Phasi $x^{TM}$  Mesh October 30, 2017 Protocol DVL-HE-011

## 6.3.1 Subjects Not Implanted and Surgical Repair Failures

Subjects who are screened but do not have the test device placed should be considered a screen failure and treated per hospital standard of care. Screen failure subjects who experience a protocol defined AE will be followed through satisfactory resolution or stabilization of the event.

Reason for failure of the surgical repair procedure, as well as all information outlined in Section 6.2.3 must be recorded in the source documentation.

## 6.3.2 Subjects Successfully Implanted

Subjects successfully implanted with Phasix<sup>TM</sup> Mesh will be followed as per the protocol defined follow-up procedures (see Table of Study Events).

#### 6.3.3 Assessments

Subjects should report to their respective study site for follow-up visits at the following times:

- 1 month assessment: Day  $30 \pm 7$  days post device placement
- 3 month assessment: Day 90 + 30 days post device placement
- 6 month assessment: Day 180 + 30 days post device placement
- 12 month assessment: Day 365 ± 30 days post device placement
- 18 month assessment: Day  $545 \pm 30$  days post device placement
- 24 month assessment: Day  $730 \pm 30$  days post device placement
- 30 month assessment: Day 910 + 30 days post device placement
- 36 month assessment: Day 1095 + 30 days post device placement
- 42 month assessment: Day 1275 + 30 days post device placement
- 48 month assessment: Day 1460 + 30 days post device placement
- 54 month assessment: Day  $1640 \pm 30$  days post device placement
- 60 month assessment: Day 1825 ± 30 days post device placement

At each study visit (see exception below for the 30, 42, and 54 month assessments) the following procedures will be completed and these data recorded in source documentation and on the eCRF:

- Physical exam to check for hernia recurrence and surgical complications. Note: If the subject undergoes imaging for any reason and a recurrent hernia is identified, it must be recorded.
- Surgical Pain Scale (VAS)
- Carolinas Comfort Scale<sup>®</sup>
- SF-12<sup>®</sup>
- Concomitant pain medication usage (all pain medication will be captured at baseline. Hernia associated pain medication only will be captured at 12,24, 36, 48, and 60 months)
- Assessment of AEs/complications

#### 6.3.3.1 Roll in Visit

The Roll in Visit should be completed in clinic where eligible subjects should be reconsented and confirmed that no abdominal surgeries were performed at the site of the index procedure. Sites with IRB approval of the extension study may complete the Roll in Visit with eligible subjects in combination with the 36 Month Follow Up visit.

6.3.3.2 30 Month Follow Up (910 days  $\pm$  30 days), 42 Month Follow Up (1275  $\pm$  30 days), 54 Month Follow Up (1640 days  $\pm$  30 days)

Phasix<sup>TM</sup> Mesh Protocol DVL-HE-011

> A telephone contact should be scheduled with the subject and completed by the Investigator. The following information will be collected:

- Symptoms suggestive of hernia recurrence
- Symptoms suggestive of surgical site infections
- Any adverse events relating to the device, procedure, or abdominal space since the last study assessment

Version 4.0

If the Investigator determines the responses provided by the subject demands a physical exam be conducted, an office visit will be scheduled. The office visit will be included as part of the 30, 42 or 54 Month Follow Up assessment (not an Unscheduled Visit) and will require all study assessments listed in Section 6.3.3 to be completed.

#### 6.3.4 **Unscheduled Visits**

If the subject has an evaluation related to the abdomen or abdominal organs at any time during the subject's study follow-up period, the subject will undergo unscheduled visit study procedures (see Table of Study Events).

## TABLE OF STUDY EVENTS

| Study Procedure | Screening<br>and Baseline<br>Period | Surgery | 1 Month<br>Visit | 3 Month<br>Visit | 6 Month<br>Visit | 12 Month<br>Visit | 18 Month<br>Visit | 24 Month<br>Visit | 30 Month<br>Visit <sup>3</sup> | 36 Month<br>Visit <sup>4</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (days) | Within 30<br>days of<br>consent | 0 | 30 <u>+</u> 7 | 90 <u>+</u> 30 | 180 <u>+</u> 30 | 365 <u>+</u> 30 | 545 <u>+</u> 30 | 730 <u>+</u> 30 | 910 <u>+</u> 30 | 1090 <u>+</u> 30 |
| Describe study to potential subject | X | | | | | | | | | |
| Obtain informed consent | X | | | | | | | | | |
| Verify eligibility criteria | X | $\mathbf{X}^{1}$ | | | | | | | | |
| Collect demographics and medical history | X | | | | | | | | | |
| Conduct physical examination | X | | X | X | X | X | X | X | | X |
| Placement Procedure of Device | | $\mathbf{X}^2$ | | | | | | | | |
| Surgical Pain Scale (VAS) | X | | X | X | X | X | X | X | | X |
| Carolinas Comfort Scale® | X | | X | X | X | X | X | X | | X |
| SF-12® | X | | X | X | X | X | X | X | | X |
| Collect adverse events/complications | | X | X | X | X | X | X | X | X | X |
| Collect pain medication usage | X | | | | | X | | X | | X |
| Schedule next follow-up visit | X | X | X | X | X | X | X | X | X | |

Intraoperative verification of hernia size

<sup>2</sup> See Section 6.2 for surgical procedure details

<sup>3</sup> Investigator will determine whether clinic visit is necessary based on subject responses. Site will complete all study procedures at clinic visit.

## 6.4 TABLE OF STUDY EVENTS (cont.)

| Study Procedure | Roll in Visit <sup>4</sup> | 42 Month<br>Visit | 48 Month<br>Visit | 54 Month<br>Visit | 60 Month<br>Visit <sup>3</sup> | Unschedule<br>d<br>Visit/Early<br>Termination |
|---|---|---|---|---|---|---|
| Visit Window (days) | Re-consent | 1275 <u>+</u> 30 | 1460 <u>+</u> 30 | 1640 <u>+</u> 30 | 1825 <u>+</u> 30 | |
| Describe study to subject | X | | | | | |
| Obtain informed consent | X | | | | | |
| Verify eligibility criteria | X | | | | | |
| Collect demographics and medical history | | | | | | |
| Conduct physical examination | X | | X | | X | X |
| Placement Procedure of Device | | | | | | |
| Surgical Pain Scale<br>(VAS) | X | | X | | X | X |
| Carolinas Comfort Scale® | X | | X | | X | X |
| SF-12® | X | | X | | X | X |
| Collect adverse events/complications | X | X | X | X | X | X |
| Collect pain medication usage | X | | X | | X | |
| Schedule next follow-up visit | X | X | X | X | | |

<sup>&</sup>lt;sup>4</sup> Roll in Visit should be completed in the clinic and may be combined with the 36 Month F/U visit

## 6.5 Withdrawal and/or Early Termination

Subjects will be informed that they have the right to withdraw from the study at any time, without affecting their future care. Subjects may also be discontinued from the study, if the Investigator determines it is in the best interest of the subject.

Additionally, subjects may be discontinued for reasons including, but not limited to the following:

- Consent is withdrawn
- Lost to follow-up (LTF)
- Death
- Investigator withdrawal of subject
- Other

A subject is considered LTF if the investigational site personnel are unable to locate the subject despite two documented attempts to notify the subject via telephone and a third attempt by certified mail.

A subject is considered an Early Termination (ET), if discontinuation occurs after successful implant of the test device. The site should attempt to bring the subject back to complete all ET visit study procedures (see Table of Study Events).

Once a subject discontinues from the study, the Investigator must complete a Study Completion eCRF and the reason for subject discontinuation must be fully documented.

## 7 STATISTICAL METHODS

This section describes the planned statistical analyses for this study. A detailed Statistical Analysis Plan (SAP) will be completed and placed on file prior to database lock. The SAP will contain a comprehensive explanation of the methodology used in the statistical analyses described below.

## 7.1 Study Hypothesis

There is no formal statistical hypothesis for this observational post-market study. The study will follow eligible, high risk patients implanted with the Phasix<sup>TM</sup> Mesh for hernia repair in order to assess long-term recurrence and surgical site infection rates.

## 7.2 Sample Size Considerations

This study is projected to enroll up to 120 subjects at approximately 16 sites. The sample size of 120 subjects is based on potential adequacy of data to meet the study objectives. It is not based on any statistical consideration.

## 7.3 Data Analysis

The Intent-to-treat (ITT) population consists of all enrolled subjects who have signed the Informed Consent Form. The modified ITT (mITT) population is defined as those subjects in the ITT population in whom Phasix Mesh has been implanted. A Per-Protocol (PP) population may be created if there are subjects who have any major protocol deviations. The PP population will consist of any subjects in the mITT population who do not have any major protocol deviation. The protocol deviations that are considered to have a "major" grade will be defined a priori in the analysis plan. All analyses will be primarily based on the mITT population. Primary analyses may be performed for PP population as well.

Demographics and baseline characteristics will be summarized using the ITT population. Summary statistics for categorical variables will include frequency counts and percentages and for continuous variables mean, standard deviation, minimum, median and maximum.

The primary endpoints of hernia recurrence rate and surgical site infection rate will be reported by visit along with their 95% confidence intervals based on the mITT population. The calculation of rates at each time point will be based on available data at the time point. Missing data will not be imputed. Additionally, a Kaplan-Meier survival analysis will be performed.

The secondary endpoints of VAS pain scale, Carolinas Comfort Scale and SF-12<sup>®</sup> will be summarized based on the mITT population with mean, standard deviation, minimum, median and maximum presented by visit. Other secondary endpoints will be summarized as appropriate.

Subjects who do not have Phasix<sup>TM</sup> Mesh implanted will have their AEs summarized separately and their outcome data will not be collected or analyzed.

Exploratory analyses on subpopulations may be performed.

#### 8 ADVERSE EVENTS

The Investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE, as provided in this protocol. All AEs that occur during the study should be treated with established standards of care that will protect the life and health of the study subjects.

AEs will be collected from the time of enrollment (AE onset after signing ICF) through the end of study participation (either study completion or early discontinuation) and will be documented in the medical record or source document and on study eCRFs. All events will be followed to satisfactory resolution or stabilization.

#### 8.1 **Definition Of Adverse Events**

In this study, an AE is defined as any undesirable clinical event occurring in the abdominal space including the lower abdominal, inguinal and pubic regions (including the skin), as well as any other undesirable clinical events judged to be related to the study device or surgical procedure regardless of anatomical region. Abnormal laboratory results are not to be considered AEs unless the results are accompanied by clinical signs or symptoms. The Investigator will assess the relationship of an AE to the study device or procedure as described in Section 8.5.

#### 8.2 **Definition of Serious Adverse Events**

An event will be classified as a serious adverse event (SAE) if it meets the definition of serious injury in the Medical Device Reporting Regulation [21 CFR 803.3] as listed below:

- results in, or contributes to, a death or serious injury;
- is life-threatening (i.e., the subject was at risk of death at the time of the event);
- requires in subject hospitalization or prolongation of existing hospitalization;
- results in persistent disability or incapacity (i.e., permanent impairment of a body function or permanent damage to a body structure);
- necessitates medical or surgical intervention to prevent one of the outcomes listed above in this definition (i.e., to preclude permanent impairment of a body function or permanent damage to a body structure)

NOTE: The term serious is not synonymous with severity, which may be used to describe the intensity of an event experienced by the subject.

## 8.3 Relationship of Adverse Event to Device/Procedure

Assess each AE for its relationship to the device (Phasix<sup>TM</sup>) or surgical procedures as follows:

• Device: This category should be restricted to AEs directly attributable to devices used as part of the study procedure.

• Procedure: This category should be restricted to AEs directly attributable to the study device surgical procedure.

Use the following categories for assigning the certainty of the relatedness:

- Definitely Related: An AE is definitely related if it is obvious, certain or there is little doubt regarding the relationship.
- Possibly Related: An AE is possibly related if it is capable of being related but relatively unlikely.
- Not Related: An AE is not related if it is determined that there is no plausible association.

## 8.4 Severity Of Adverse Events

Each AE should be assessed for its severity, or the intensity of an event, experienced by the subject.

- Mild: Awareness of a sign or symptom that does not interfere with the subject's activity or is transient and is resolved without treatment or sequelae.
- Moderate: May interfere with the subject's activity and require additional intervention and/or treatment, and may have additional sequelae.
- Severe: Significant discomfort to the subject and/or interferes with the subject's
  activity. Additional intervention and/or treatment are necessary. Additional sequelae
  occur. Severe is used to describe the intensity of an event experienced by the subject.

## 8.5 Reporting Of Adverse Events

If an AE occurs, all sections of the appropriate eCRF must be completed.

All Investigator-judged device- or procedure-related AEs that occur (whether serious or not) must be reported to Davol Inc. Field Assurance using the contact information provided in Section 9, within 24 hours of becoming aware of the event.

Additionally, all SAEs (whether device- or procedure-related or not) must be reported to the Sponsor within 24 hours of becoming aware of the event.

**Version 4.0** October 30, 2017

It is the responsibility of the Investigator to inform the Institutional Review Board (IRB) of AEs according to IRB requirements. The Sponsor will report to the Food and Drug Administration (FDA) as appropriate after becoming aware of a reportable event.

## 9 MECHANICAL FAILURES, MALFUNCTIONS AND DEFECTS

The Investigator will record if the surgical mesh device used in the study procedure failed to meet its performance specifications whether due to mechanical failure, malfunction or defects. This applies to: devices used in the subject, devices in which the package was opened but the device was not used for implantation in the subject, or devices with which implantation was attempted, but the device did not remain (was not used) in the subject.

A recurrence (unless it is in a different location than the study hernia) is considered a device failure if the recurrence is clearly device related, and not procedure related or an issue of patient mismanagement (e.g., use of a Vacuum Assisted Closure (VAC) system for too long; mesh used was too small to adequately cover the defect), as determined by the Investigator.

All mechanical failures, malfunctions, missing components, foreign matter inclusion or any other defects of the study device or any components of the device kit that do not perform to specifications must be promptly reported to the Davol Field Assurance Department:

Field Assurance Department

e-mail: Davol.FieldAssurance@crbard.com

Telephone: 800-556-6756 Sarah Hardy – Ext 8422

e-mail: Sarah.Hardy@crbard.com

The event must also be documented on the Device Failure eCRF and the malfunctioning device promptly returned to the manufacturer.

#### 10 CASE REPORT FORMS

The Investigator is responsible for ensuring the accuracy and completeness of all study documentation. All clinical study data will be recorded in the eCRFs provided to the investigational site.

#### 11 RISK/BENEFIT ANALYSIS

Subjects participating in this study will require hernia repair surgery as part of their standard of care. The device utilized in this study is commercially available, has 510(k) clearance from the US FDA and will be used in accordance with the indications in labeling which are in effect during the study period. This study will not pose any additional potential risk to the

health, safety, or welfare of the subject. The risks associated with hernia repair and Phasix<sup>TM</sup> Mesh are described in full in the IFUs (Appendix 2).

There is no immediate benefit to the subject for participation in this study. Collection and analysis of the data generated in this study may be of benefit to future subjects who require hernia repair.

## 12 ADMINISTRATIVE REQUIREMENTS

This study will be conducted in accordance with the Declaration of Helsinki, HIPAA requirements, Good Clinical Practices (GCP), and applicable FDA regulations (21 CFR parts 50, 54, 56 and will be exempt from the requirements of 21 CFR part 812, as per 21 CFR part 812.2(c)(2), as the device has been cleared by the FDA for commerce and will be used as per the IFU.)

### 12.1 **Publication Policy**

At the conclusion of the study, a multi-center article may be prepared for publication in a scientific journal. The publication of the principal results from any single-center experience within the study is not allowed until the preparation and publication of the multi-center results. Exceptions to this rule require the prior approval of Davol. The analysis of other prespecified and non-pre-specified endpoints will be performed by Davol or its designee. Such analyses, as well as other proposed investigations will require the approval of Davol. Davol anticipates the possibility of secondary manuscripts with principal authorship. For purposes of timely abstract presentation and publication, such secondary publications will be delegated to the appropriate principal authors, and final analyses and manuscript review for all multi-center data will require the approval of Davol.

## 12.2 Investigator Selection

The Investigator must be of good standing as an Investigator and knowledgeable in relevant areas of clinical research to ensure adherence to the requirements of the protocol, including the protection of human subjects. Other site personnel must have appropriate research experience and infrastructure to ensure adherence to the protocol and enrollment of sufficient numbers of evaluable subjects. The curriculum vitae (CV) of the Investigator will be maintained in the Sponsor files as documentation of previous medical training, and federal databases will be searched to ensure that the Investigator and/or the site are not prohibited from engaging in federally Sponsored clinical research. The Principal Investigator will sign the signature page of this protocol, agreeing to comply with all applicable government regulations and the requirements of this study.

## 12.3 Regulatory and Ethical Considerations

## 12.3.1 Institutional Review Board Approval

Before commencement of the study, the Investigator must provide Sponsor with written documentation of IRB approval. This approval must refer to the ICF and the study by both the title and the protocol number assigned by Sponsor. The Investigator, if a member of the IRB, is not to participate in the approval decision for this study. This non-participation should be noted in the approval letter.

The IRB must give written renewal of the original approval at least annually to continue the study. A copy of the written renewal must be provided to Sponsor.

## 12.3.2 Informed Consent and HIPAA Authorization

Prior to the procedure, the Investigator (or designee) must explain to each subject (or the subject's legally authorized representative) in layman's terms, the nature of the study, its purpose, expected duration, and the benefits and risks of study participation. Also, subjects will be informed of uses and disclosures of their medical information for research purposes and their rights to access information about them. The subjects must be informed of their rights to withdraw from the study at any time for any reason without sanction, penalty, or loss of benefits to which they are otherwise entitled, and that withdrawal from the study will not jeopardize their future medical care. After this explanation and before entering the study, the subject (or legally authorized representative) must voluntarily sign and date the IRB-approved ICF and HIPAA Consent Form in accordance with 21 CFR Parts 50 and 56. The subject will receive a copy of their ICF and HIPAA Consent Form.

## 12.3.3 Confidentiality

All information and data sent to Davol, Inc. or an authorized designee concerning subjects or their participation in the study will be considered confidential. All data used in the analysis and reporting of this study will be used in a manner without identifiable reference to the subject. The Investigator consents to visits by personnel of Davol, Inc. and its affiliates or designees, as well as, FDA representatives.

### 12.4 Protocol Adherence and Deviations

The study will be conducted as described in this protocol. Investigators are not permitted to deviate from this protocol except to protect patient rights, safety or well-being. Any deviations from this protocol must be documented by the Investigator. If an emergency situation arises in which the rights, safety and well-being of a subject may require immediate alternative intervention, the Investigator should act in the best interest of the subject. Sponsor and the site's IRB must be notified immediately if this occurs. This should be followed with written confirmation that describes the emergency action and outcomes, to Sponsor and per IRB reporting requirements. Protocol deviations will be reviewed during routine monitoring visits. Investigators will be required to identify preventive and corrective

actions to prevent further deviations. An Investigator may be disqualified from the study for repeated and/or egregious protocol deviations.

This protocol may be amended as necessary by the Sponsor. Any protocol amendments will be documented via an incremented version of this protocol (with relevant revision history) and a "was/is" comparison table to highlight the protocol changes. Amendments to the protocol must undergo the same approval process by the Sponsor, Investigators, IRBs and regulatory authorities as the original protocol.

## 12.5 Device Accountability

Only commercially available surgical mesh products will be used. Device accountability will not be required.

#### 12.6 **Data Collection**

The Investigator is responsible for completely and accurately recording study data in the appropriate sections of the eCRFs provided by Sponsor. The eCRFs must be signed by the Investigator or by his/her documented designee.

The Investigator is also responsible for making source documents and forms readily available for a thorough review by the study monitor at each monitoring visit. The monitor will ensure the accuracy of data recording at each investigational site by comparison to supporting source documents during periodic site visits. Adherence to proper recording of information as well as assuring that corrections are being made will also be addressed during these periodic visits.

## 12.7 Subject Compensation

To compensate subjects for their time and participation, they may receive stipends upon completion of each of the protocol specified study visits. If the subject does not complete a visit, they will not be compensated for that visit.

## 12.8 Communications with the Sponsor

Although the Investigator and his/her staff may have contact with other key individuals at the Sponsor throughout the course of the study, all communications regarding conduct of the study must be channeled through the Sponsor's clinical affairs personnel or their designees.

## 12.9 Required Documentation

An Investigator may not screen or enroll subjects until authorized to do so by the Sponsor. At a minimum, the following documentation must be received by the Sponsor prior to study commencement:

- CVs and medical licenses for the principal Investigator and sub-Investigators;
- Signed Clinical Study Agreement;
- Signed Nondisclosure Agreement;
- Signed "Protocol Signature Page" (page ii of this protocol);
- Written approval from the IRB of both the protocol and ICF;
- Signed Financial Disclosure Statement; and
- IRB Assurance of Compliance Form or equivalent.

## 13 SITE MONITORING

The study monitors are designated as agents of the Sponsor and are assigned to oversee the conduct and progress of the study and to be the principal communication link between the Sponsor and the Investigator.

The study monitors will be involved in Investigator selection and training, assurance of IRB approvals, and periodic on-site inspection and monitoring of sites and records, to ensure continued compliance with the protocol and adequacy of the Investigator and the facility to carry out the study. In addition, the monitor will verify that the device is being used in accordance with the protocol instructions.

The site may also be subject to a quality assurance audit by personnel of the Sponsor as well as by FDA representatives.

The monitor will perform several types of site visits during the course of the study. In all cases, the study monitor will provide a written summary of the visit, including necessary follow-up items, to the Investigator and Sponsor.

It is important that the Investigator(s) and the relevant site personnel are available during the monitoring visits, and possible audit, and that sufficient time is devoted to the process.

## 13.1 Study Initiation Visit

Before the study begins, the study monitor will visit the site. The purpose of this visit is to review with the Investigator and staff the provisions and proper conduct of the clinical evaluation. This includes a detailed review of the protocol and eCRFs with instructions as to their completion, as well as reviewing regulations pertaining to the conduct of the clinical study. Arrangement for timely and accurate reporting of clinical data and relevant medical events will be established as well as ensuring safe and secure storage for the study devices.

The study monitor will:

- Confirm that the ICF to be used is the one approved by the IRB;
- Verify that all necessary documents are on file at the site; and
- Confirm that there are provisions to continue and maintain all documents and records throughout the study as required by GCP regulations.

## 13.2 Ongoing Monitoring Visits

The study monitor will maintain personal contact with the Investigator and staff throughout the study by telephone, e-mail, fax, mail, and on-site visits. On-site monitoring will begin after the first subjects are enrolled and continue until the study is completed. The monitoring will assure continued protocol compliance, adequate subject enrollment, accurate data reporting (including the comparison of eCRFs with subject records), device accountability (if required), and continued IRB acceptance of the study. The study monitor will evaluate and summarize the results of each visit in written reports, identifying any ongoing data problems with any study site and specifying recommendations for resolution of noted deficiencies. A formal monitoring plan will describe the planned extent of source data verification.

## 13.3 Final Monitoring Visit

At the completion of the study, the study monitor will conduct a final on-site visit. The purpose of this visit is to collect all outstanding study data documents, confirm that the Investigator's files are accurate and complete, review the record retention requirements with the Investigator, provide the return of unused devices (if required) to the sponsor, review records which account for device shipment (if required), and assure that all applicable requirements for closure of the study are met. The actions and observations made at this visit will be recorded and filed.

#### 14 TERMINATION OF STUDY

Sponsor reserves the right to suspend enrollment or terminate the study at any time as set forth in the Clinical Study Agreement. Written notice will be submitted to the Investigator in advance of such termination.

Sponsor may suspend enrollment or terminate the study at a specific site for reasons including, but not limited to, inadequate data collection, low subject enrollment rate, achievement of the total enrollment, or non-compliance with the protocol or other clinical research requirements.

## 15 REPORTING REQUIREMENTS

The Investigator must promptly report to Sponsor any withdrawal of IRB approval at the site. Additional reporting requirements of the Investigator include:

- Reporting all ICF violations to the IRB
- Reporting all device related AEs to Davol Field Assurance Department

## 16 RECORD RETENTION

The investigator shall retain all study records for a period of 2 years after the investigation is terminated or completed, or until the records are no longer required as determined by the Sponsor. The investigator may withdraw from the responsibility to maintain records for the period required and transfer custody of the records to any other person who will accept responsibility for retaining them with pre-approval. Notice of a transfer shall be given to the Sponsor not later than 10 working days after transfer occurs.

Version 4.0

## 17 REFERENCES

- 1. Cobb W, Kercherk, Heniford B. Laproscopic repair of incisional hernias. The Surgical Clinics of North America 2005;85: 91 103.
- 2. Mudge M, Hughes LE. Incisional hernia: a 10-year prospective study of incidence and attitudes. Br J Surg 1985;72: 70 71.
- 3. Luijendijk R. Hop E, van den Tol M, et al. Comparison of surgical repair with mesh repair for incisional hernia. New Engl J Med 2000;343: 392 398.
- 4. Anthony T, Bergen PC, Kim L, et al. Factors affecting recurrent following incisional herniorrhaphy. World J of Surg 2000;24: 95 101.
- 5. Burger J, Luijendijk R, Hop W, et al. Long-term follow-up of a randomized controlled trial of suture versus mesh repair incisional hernia. Ann Surg 204;240: 578 583.
- 6. van Geffen H, Simmermacher R, van Vroonhoven T, van der Werken C. Surgical treatment of large contaminated abdominal wall defects. J Am Coll Surg 2005;201: 206 212.
- 7. George C, Ellis H. The results of incisional hernia: a twelve-year review. Ann R Coll Surg Engl 1986; 68:185-187.
- 8. Ramirez RM, Ruas E, Dellon AL. "Components separation method for closure of abdominal-wall defects: An anatomic and clinical study. Plast Reconstruct Surg 1990; 86:519 526.
- 9. DiBello J, Moore J. Sliding myofascial flap of the rectus abdominis muscle for the closure of recurrent ventral hernias. Past Reconstr Surg 1996; 98:464 469.
- 10. Girotto J, Ko M, Redett, et al. Closure of chronic abdominal wall defects: a long-term evaluation of the component separation method. Ann Plat Surg 1999; 42:385 395.
- 11. Shestak K, Edington H, Johnson R. The separation of anatomical components technique for the reconstruction of massive midline abdominal wall defects: anatomy, surgical technique, application and limitations revisited. Plast Reconstr Surg 2000; 105:731-738.
- 12. Lowe J, Garza J, Bowman J, et al. Endoscopically assisted "components separation technique" for closure of abdominal wall defects. Plat Reconstr Surg 2000; 105:720 729.

- 13. Markar SR, Karthikesalingam A, Alam F, Tang TY, Walsh SR, Sadat U. Partially or completely absorbable versus nonabsorbable mesh repair for inguinal hernia: a systematic review and meta-analysis. Surg Laparosc Endosc Percutan Tech. 2010 Aug; 20(4):213-9. Review. PubMed PMID: 20729687.
- 14. Hakeem A, Shanmugam V. Inguinodynia following Lichtenstein tension-free hernia repair: A review. World J Gastroenterol. 2011;17(14):1791-1796.
- 15. Sadowski B, Rodriguez J, Symmonds R, Roberts J, Song J, Rajab MH, Cummings C, Hodges B; The Scott and White Outcomes and Effectiveness Registry Group. Comparison of polypropylene versus polyester mesh in the Lichtenstein hernia repair with respect to chronic pain and discomfort. Hernia. Published online: 14 July 2011. Doi: 10.1007/s10029-011-0841-x.
- 16. Martin DP, Williams SF. Medical applications of poly-4-hydroxybutyrate: a strong flexible absorbable biomaterial. Biochemical Engineering Journal 2003;16:97-105.
- 17. Chen GQ, Wu Q. The application of polyhydroxyalkanoates as tissue engineering materials. Biomaterials. 2005 Nov26;33:6565-78.
- 18. Wu Q, Wang Y, Chen GQ. Medical application of Microbial Biopolyesters Polyhydroxyalkanoates. Artificial Cells, Blood Substitutes, and Biotechnology 2009;37:1-12.
- 19. Martin DP, Badhwar A, Shah DV, Rizk S, Eldridge SN, Gagne DH, Ganatra A, Darois RE, Williams SF, Tai HC, Scott JR. Characterization of poly-4-hydroxybutyrate mesh for hernia repair applications. Journal of Surgical Research. 2013 Apr 2; Epub ahead of print.
- 20. Deeken C, Matthews BD. Characterization of the Mechanical Strength, Resorption Properties, and Histologic Characteristics of a Fully Absorbable Material (Poly-4-Hydroxybutyrate PHASIXTM Mesh) in a Porcine Model of Hernia Repair. ISRN Surgery. 2013 Apr 23;2013:1-12.
- 21. Data on file. Warwick, RI, USA: Davol Inc., RPT3803626, Rev 0.
- 22. Albertsmeier M, Seiler CM, Fischer L, Baumann P, Husing J, Seidlmayer C., Franck A, Jauch KW, Knaebel HP, Buchler MW. Evaluation of the safety and efficacy of MomoMax suture material for abdominal wall closure after primary midline laparotomy a controlled prospective multicenter trial. Langenbecks Arch Surg. 2012 Mar; 397(3):363-71)
- 23. Morris PJ, Malt RA. Oxford textbook of Surgery Volume 1. Oxford: Oxford Medical Publications, Oxford University Press, 1994.

Davol Inc. Version 4.0 Phasi $x^{TM}$  Mesh October 30, 2017 Protocol DVL-HE-011

24. Mangram AA, Horan TC, Peron ML, Silver LC, Jarvis WR. Guidance for prevention of surgical site infection, 1999. Infection Control and Hospital Epidemiology. 1999;

25. CDC Surgical Site Infection (SSI) Event Protocol http://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf

20(4):247 - 278.

Davol Inc. Version 4.0 Phasi $x^{TM}$  Mesh October 30, 2017 Protocol DVL-HE-011

## 18 APPENDICES

## **Appendix 1: Principal Investigator Information**

John Scott Roth, MD University of Kentucky Medical Center 800 Rose Street, #C222 Lexington, Kentucky 40536

Phone: 859-323-6346 ext. 232

Appendix 2: Phasix<sup>TM</sup> Mesh Instructions for Use



# INSTRUCTIONS FOR USE









Distributed by: Davol Inc. Subsidiary of C. R. Bard, Inc. 100 Crossings Boulevard Warwick, RI 02886 USA 1-401-825-8300 1-800-556-6275

Medical Services & Support Clinical Information Line 1-800-562-0027

Manufactured by: Tepha, Inc. 99 Hayden Avenue, Suite 360 Lexington, MA 02421 USA



#### PRODUCT DESCRIPTION

PHASIX<sup>™</sup> Mesh is a resorbable mesh prepared from poly-4-hydroxybutyrate (P4HB). P4HB is produced from a naturally occurring monomer and is processed into monofilament fibers and knitted into a surgical mesh.

Phasix™ Mesh degrades through a process of hydrolysis and a hydrolytic enzymatic digestive process. It has been developed to minimize the variability of resorption rate (loss of mass) and strength and provide support throughout the expected period of healing.

Pre-clinical implantation studies indicate that the resorption of the Phasix™ fibers is minimal throughout the 12 week expected period of healing and up to about 26 weeks post implantation. Resorption of the fibers is essentially complete in 12 to 18 months.

#### INDICATIONS

Phasix™ Mesh is indicated to reinforce soft tissue where weakness exists, such as the repair of hernia or other fascial defects that require the addition of a reinforcing or bridging material to obtain the desired surgical result.

#### CONTRAINDICATIONS

Because Phasix<sup>™</sup> Mesh is fully resorbable, it should not be used in repairs where permanent wound or organ support from the mesh is required.

#### WARNINGS

- Device manufacture involves exposure to tetracycline hydrochloride and kanamycin sulfate. The safety and product use for patients with hypersensitivities to these antibiotics is unknown. Use of this device in patients with known allergies to tetracycline hydrochloride or kanamycin sulfate should be avoided.
- 2. The safety and effectiveness of Phasix™ Mesh in neural tissue and in cardiovascular tissue has not been evaluated or established.
- 3. The safety and effectiveness of Phasix™ Mesh in pediatric use has not been evaluated or established.
- The placement of Phasix™ Mesh in direct contact with bowel or viscera is not recommended.
- If an infection develops, treat the infection aggressively. Consideration should be given regarding the removal of the mesh. An unresolved infection may require removal of the device.
- This device is supplied sterile. Inspect the device and packaging prior to use to be sure they are intact and undamaged.
- 7. This device is for single use only. Do not resterilize or reuse any portion of the Phasix™ Mesh.
- If unused prosthesis has been in contact with instruments or supplies used on a patient or contaminated with body fluids, discard with care to prevent risk of transmission of viral infections.

#### PRECAUTIONS

- Please read all instructions prior to use.
- Only physicians qualified in the appropriate surgical techniques should use this device. Users should be familiar with strength and mesh size requirements. Improper selection, placement, positioning and fixation of the devices can cause subsequent undesirable results.

#### ADVERSE REACTIONS

In pre-clinical testing, Phasix™ Mesh elicited a minimal tissue reaction characteristic of foreign body response to a substance. The tissue reaction resolved as the mesh was resorbed. Possible complications include infection, seroma, pain, mesh migration, wound dehiscence, hemorrhage, adhesions, hematoma, inflammation, extrusion and recurrence of the hernia or soft tissue defect.

#### DIRECTIONS FOR USE

Phasix™ Mesh may be cut to shape or size desired for each specific application. To prevent recurrences when repairing hernias, a mesh larger than the defect is required to ensure adequate coverage. The mesh is to be positioned so its edges extend beyond the margins of the defect.

It is recommended that surgical fixation be placed  $\frac{1}{4}$  to  $\frac{1}{2}$  inches (6 to 12mm) apart at a distance approximately  $\frac{1}{4}$  inch (6mm) from the edge of the mesh. The edges are then fixated to assure proper closure under correct tension.

#### HOW SUPPLIED

Phasix™ Mesh is available in single packets as a sterile, undyed fabric mesh in single sheet sizes of varying widths and lengths.

#### STORAGE

Store at room temperature. Avoid prolonged exposure to elevated temperatures. The indicator should be white or light grey. If the indicator is black on the box, check the indicator on the foil pouch. If the indicator is black on the foil pouch, do not use the product.

#### TRACEABILITY

A traceability label that identifies the type, size, expiration date and lot number of the device is attached to every package. This label should be affixed to the patient's permanent medical record to clearly identify the device that was implanted.

Copyright © 2010 C. R. Bard, Inc. All Rights Reserved.

**Bard**, **Davol** and **Phasix** are trademarks and/or registered trademarks of C. R. Bard, Inc. or an affiliate.

## **Appendix 3: Surgical Site Infection Classification**<sup>24</sup>

Superficial Incisional Surgical Site Infections (SSI)

Infection occurs within 30 days after the operation and

Infection involves only the skin or subcutaneous tissue around the incision and at least one of the following:

- 1. Purulent drainage with or without laboratory confirmation, from the superficial incision.
- 2. Organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision.
- 3. At least one of the following signs or symptoms of infection: pain or tenderness, localized swelling, redness or heat and superficial incision is deliberately opened by a surgeon, unless the culture is negative.
- 4. Diagnosis of superficial incisional SSI by the surgeon or attending physician.

NOTE: Do not report the following as SSI:

- 1. Stitch abscesses (minimal inflammation and discharge confined to the points of suture penetration)
- 2. Infection of the episiotomy or neonatal circumcision sites
- 3. Infected burn wound.
- 4. Incisional SSI that extends into the fascial and muscle layers (see definition for Deep Incisional Surgical Site Infections below).

Note: Specific criteria are used for identifying infected episiotomy and circumcision sites and burn wounds.

#### Deep Incisional SSI

Infection occurs within 30 days after the operation if no implant is left in place or within one year if implant is in place and the infection appears to be related to the operation. and

Infection involves deep soft tissues (e.g., fascia and muscle layers) of the incision and at least one of the following:

- 1. Purulent drainage from the deep incision but not from the organ/space of the surgical site.
- 2. A deep incision spontaneously dehisces or is deliberately opened by a surgeon when the patient has at least one of the following signs: fever (>38°C), localized pain or tenderness unless the culture is negative.
- 3. An abscess or other evidence of infection involving the deep incision is found on direct examination, during reoperation, or by histopathologic or radiologic examination.
- 4. Diagnosis of a deep SSI by a surgeon or attending physician.

### Notes:

- 1. Report infection that involves both superficial and deep incision as deep incisional SSI.
- 2. Report an organ / space SSI that drains through the incision as deep incisional SSI.

# **Appendix 4: Surgical Wound Classification**<sup>25</sup>

- Class I/Clean: An uninfected operative wound in which no inflammation is encountered and the respiratory, alimentary, genital, or uninfected urinary tract is not entered. In addition, clean wounds are primarily closed and, if necessary, drained with closed drainage. Operative incisional wounds that follow nonpenetrating (blunt) trauma should be included in this category if they meet the criteria.
- Class II/Clean-Contaminated\*: An operative wound in which the respiratory, alimentary, genital, or urinary tracts are entered under controlled conditions and without unusual contamination. Specifically, operations involving the biliary tract, appendix, vagina, and oropharynx are included in this category, provided no evidence of infection or major break in technique is encountered.
- Class III/Contaminated\*: Open, fresh, accidental wounds. In addition, operations with major breaks in sterile technique (e.g., open cardiac massage) or gross spillage from the gastrointestinal tract, and incisions in which acute, non-purulent inflammation is encountered including necrotic tissue without evidence of purulent drainage (e.g. dry gangrene) are included in this category.
- Class IV/Dirty-Infected\*: Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera. This definition suggests that the organisms causing postoperative infection were present in the operative field before the operation.

<sup>\*</sup> NOTE: In this study, subjects with Class II, Class III and Class IV wounds are to be excluded from enrollment.